CLINICAL TRIAL: NCT04513457
Title: Perioperative Chemotherapy Versus Surgery for Resectable Colorectal Liver Metastases: a Multicenter Propensity Score Matched Analysis on Long-term Outcomes
Brief Title: Chemotherapy for Resectable Colorectal Liver Metastases
Status: Completed | Type: Observational
Sponsor: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Collaborators: Marcello Di Martino (Unknown)
Responsible Party: Sponsor
Other Study IDs: Chemotherapy-liver-metastases
Record Dates: First submitted 2020-08-11; First posted 2020-08-14 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Metastatic Colorectal Cancer; Metastatic Liver Cancer
Keywords: Colorectal liver metastases; Liver resection; Hepatectomy
MeSH Terms: conditions — Colorectal Neoplasms; Liver Neoplasms | interventions — Hepatectomy; Neoadjuvant Therapy; Chemotherapy, Adjuvant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Liver resection and Neoadjuvant chemotherapy: Liver resection and Neoadjuvant chemotherapy
  Interventions: Other: Liver resection and Neoadjuvant chemotherapy
- Liver resection and Adjuvant chemotherapy: Liver resection and Adjuvant chemotherapy
  Interventions: Other: Liver resection and Adjuvant chemotherapy
- Liver resection, Neoadjuvant and Adjuvant chemotherapy: Liver resection, Neoadjuvant chemotherapy and Adjuvant chemotherapy
  Interventions: Other: Liver resection, Neoadjuvant chemotherapy and Adjuvant chemotherapy
- Liver resection: Liver resection
  Interventions: Procedure: Liver resection

INTERVENTIONS:
Other: Liver resection and Neoadjuvant chemotherapy
  Groups: Liver resection and Neoadjuvant chemotherapy
Other: Liver resection and Adjuvant chemotherapy
  Groups: Liver resection and Adjuvant chemotherapy
Other: Liver resection, Neoadjuvant chemotherapy and Adjuvant chemotherapy
  Groups: Liver resection, Neoadjuvant and Adjuvant chemotherapy
Procedure: Liver resection
  Groups: Liver resection

SUMMARY:
There is a degree of uncertainty regarding the role of perioperative chemotherapy (CTx) in the treatment of resectable colorectal liver metastases (CRLM). In the clinical practice, the combination of surgery and CTx is increasingly accepted as treatment for CRLM, especially in the context of patients with synchronous disease or metachronous disease with a high risk of recurrence. However, controversy exists whether all patients with resectable CRLM benefit from perioperative CTx.

There is paucity of good quality studies on this topic. A pooled analysis of two phase III randomized clinical trial, closed prematurely because of slow accrual, showed a marginal statistical significance in favor of adjuvant CTx. Nevertheless, long term results of the EPOC trial founded benefit in disease free survival (DFS) with no difference in overall survival (OS) when perioperative CTx with FOLFOX4 was compared with surgery alone for resectable CRLM. Furthermore, a retrospective series from Ayez et al showed that patients with a high CRS benefit from neo-adjuvant CTx while in patients with a low risk profile did not. On the other side, another retrospective series from the MSKCC showed the timing of additional CTx for resectable CRLM was not associated with improved outcomes. The ongoing CHARISMA trial is currently comparing the outcomes of neo-adjuvant CTx followed by surgery versus surgery alone in high-risk patients with resectable CRLM.

This uncertainty regarding CRLM management may partly be due to the fact that these studies are not well powered to detect minor differences in long term outcomes and they often involved a very heterogenous group of patients with both synchronous and metachronous CRLM, not stratified by clinical risk score (CRS) as described by Fong et al.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years with resectable liver metastases of histologically confirmed primary colorectal carcinoma.
* Minimum follow-up of five years.

Exclusion Criteria:

* Patients with extrahepatic disease

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients undergoing liver resection for colorectal metastases between January 1, 2010 and December 31, 2014, inclusive
Sampling Method: Non-Probability Sample
Enrollment: 967 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Overall survival based on perioperative treatment | 5 years of follow-up
  Overall survival based on perioperative treatment
Cancer survival based on perioperative treatment | 5 years of follow-up
  Cancer survival based on perioperative treatment
Disease-free survival based on perioperative treatment | 5 years of follow-up
  Disease-free survival based on perioperative treatment
Peri-operative morbidity | 5 years of follow-up
  Peri-operative morbidity
Peri-operative mortality | 5 years of follow-up
  Peri-operative mortality

SECONDARY OUTCOMES:
Overall survival, cancer survival and disease-free survival related with biological markers | 5 years of follow-up
  Overall survival, cancer survival and disease-free survival related with biological markers
Overall survival, cancer survival and disease-free survival related with hidden no resected liver lesions. | 5 years of follow-up
  Overall survival, cancer survival and disease-free survival related with hidden no resected liver lesions.
Overall survival, cancer survival and disease-free survival based related with simultaneous thermal ablation performed at the same time of the surgical excision. | 5 years of follow-up
  Overall survival, cancer survival and disease-free survival based related with simultaneous thermal ablation performed at the same time of the surgical excision.

CONTACTS AND LOCATIONS:
Locations (9):
- Centre Hospitalier Universitaire de Reims, Reims, France
- Spain (7):
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Clínico Universitario de Valencia, Valencia, Valencia
  - Hospital Universitario de Badajoz, Badajoz
  - Hospital Dr. Josep Trueta, Girona
  - Hospital Universitario de Jaén, Jaén
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
- Liverpool University Hospitals NHS Foundation Trust, Liverpool, United Kingdom